CLINICAL TRIAL: NCT01294020
Title: A Phase II, Open-Label, Multi-Center Study to Compare the Pharmacokinetics of Tacrolimus in Stable Pediatric Allograft Recipients Converted From a Prograf® Based Immunosuppressive Regimen to a Tacrolimus Prolonged Release, Advagraf® Based Immunosuppressive Regimen, Including a Long-Term Follow-Up
Brief Title: Study to Compare the Pharmacokinetics of Tacrolimus in Stable Pediatric Allograft Recipients Converted From Prograf® to Advagraf®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PMR-EC-1206; 2010-020925-42 (EudraCT Number); 2024-517571-20-00 (Registry Identifier: CTIS(EU))
Record Dates: First submitted 2011-02-03; First posted 2011-02-11 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Intestine Transplantation; Kidney Transplantation; Lung Transplantation; Liver Transplantation; Heart Transplantation
Keywords: Transplant; Liver; Tacrolimus; Kidney; Heart; Lung; Immunosuppression; Advagraf; Pharmacokinetics
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tacrolimus Prolonged Release (Experimental): Participants receive tacrolimus prolonged release once daily starting from day 1 for 4 weeks for in Part A, and continue to receive tacrolimus prolonged release once daily up to end of Part B of the study.
  Interventions: Drug: Tacrolimus; Drug: Tacrolimus prolonged release

INTERVENTIONS:
Drug: Tacrolimus — Oral capsule
  Other Names: Prograf; FK506
Drug: Tacrolimus prolonged release — Oral capsule
  Other Names: FK506E; MR4; Advagraf; tacrolimus modified release; Astagraf XL; Graceptor; Prograf XL

SUMMARY:
Parts A & B: Conversion of stable pediatric allograft recipients from Prograf® immunosuppression to Advagraf® immunosuppression to compare exposure and one year follow-up for safety and efficacy.

Part C: Continuation of long-term follow-up and provision of ongoing study medication to subjects to whom Advagraf® is currently not available.

DETAILED DESCRIPTION:
Part A: On Day 1 subjects will be converted from their routine Prograf®-based immunosuppressive regimen to a Prograf®-based immunosuppressive regimen supplied by the Sponsor as study medication and continue treatment until Day 7. The daily dose of the study medication must be the same [1:1 (mg:mg)] as the Prograf® dose received during the 30-day screening period.

On Day 7 the first 24 hour PK profile will be started. Samples will be taken over a 24 hour period and will be completed on Day 8.

On Day 8 subjects will be switched to once-daily Advagraf® on a 1:1 (mg:mg) total daily dose basis and continue treatment until Day 14.

On Day 14 the second 24-hour PK profile will be started. Samples will be taken over a 24-hour period and will be completed on Day 15.

Part B: One year follow-up period to evaluate safety and efficacy of tacrolimus when administered as an Advagraf®-based immunosuppressive regimen.

Part C: Continuation of long-term follow-up (from Day 365 onwards). Patients who have completed Part B and to whom continued treatment with Advagraf® is not currently available, will be offered participation in a continuation of long-term follow-up (Part C). Part C will continue until Advagraf® becomes available to these patients or these patients' discontinuation, whichever is the earliest.

Part C applies to patients in the following countries: United Kingdom, Czech Republic, Germany, Italy, and Poland only.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to swallow intact study medication capsules
* Received a single solid organ transplant at least 6 months prior to entry into the study
* The subject's parent(s), or their legal representative(s), has been fully informed and has given written informed consent to participate in the study. The subject has given assent where applicable
* Has been receiving a Prograf® based immunosuppressive regimen for a minimum of 3 months
* Negative pregnancy test prior to enrolment (females)
* Must agree to practice effective birth control during the study
* Stable whole blood trough levels of tacrolimus in the range of 3.5 - 15ng/mL (+/-0.5ng/mL) and clinically stable in the opinion of the Investigator

Exclusion Criteria:

* Previously received a multiple organ transplant
* Any rejection episode within 3 months prior to enrolment or within the last 6 months that required anti-lymphocyte antibody therapy, or 2 or more rejection episodes within the last 12 months
* Currently receiving Rapamycin, Certican or MPA (Myfortic®)
* Chronic dysfunction of the allograft, in the opinion of the Investigator
* Major changes in their immunosuppressive regimen within the last 3 months prior to entry into the study
* The subject is pregnant or breast feeding

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2011-05-25 (Actual); Primary Completion 2015-10-25 (Actual); Study Completion 2025-11-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-time Curve from Time 0 to Time 24 Hours (AUC0-24h) for Tacrolimus and Tacrolimus Prolonged Release | Day 7 (for tacrolimus) and day 14 (for tacrolimus prolonged release) at predose and 1, 2, 4, 6, 12, 13, 14, 16, 18 and 24 hours postdose

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of Tacrolimus and Tacrolimus Prolonged Release | Day 7 (for tacrolimus) and day 14 (for tacrolimus prolonged release) at predose and 1, 2, 4, 6, 12, 13, 14, 16, 18 and 24 hours postdose
Time to Attain Maximum Concentration (tmax) of Tacrolimus and Tacrolimus Prolonged Release | Day 7 (for tacrolimus) and day 14 (for tacrolimus prolonged release) at predose and 1, 2, 4, 6, 12, 13, 14, 16, 18 and 24 hours postdose
Trough Concentration (C24) for Tacrolimus and Tacrolimus Prolonged Release | Days 7 and 14, 24 hours after dosing
Number of Participants with Acute Rejections | Up to Week 54
  Rejection episodes/acute rejections are indicated by clinical and/or laboratory signs, and are classified according to their rejection specific treatment: •Spontaneously Resolving Acute Rejection: not treated with new or increased corticosteroid medication, antibodies or any other medication and resolved, irrespective of any tacrolimus dose changes; •Corticosteroid Sensitive Acute Rejection: treated with new or increased corticosteroid medication only and which has resolved, irrespective of any tacrolimus dose changes; •Corticosteroid Resistant Acute Rejection: did not resolve following treatment with corticosteroids; - Resolved with further treatment: any acute rejection with an end date AND a treatment other than corticosteroid used; - Unresolved with further treatment: any acute rejection with no end date AND a treatment other than corticosteroid used; - Unresolved with no further treatment: any acute rejection with no end date AND ONLY corticosteroid treatment was used.
Number of Participants with Biopsy Proven Acute Rejections (BPARs) | Up to Week 54
  BPAR episodes are defined as acute rejection episodes confirmed by biopsy, and are classified according to their rejection specific treatment: •Spontaneously Resolving Acute Rejection: not treated with new or increased corticosteroid medication, antibodies or any other medication and resolved, irrespective of any tacrolimus dose changes; •Corticosteroid Sensitive Acute Rejection: treated with new or increased corticosteroid medication only and which has resolved, irrespective of any tacrolimus dose changes; •Corticosteroid Resistant Acute Rejection: did not resolve following treatment with corticosteroids; - Resolved with further treatment: any acute rejection with an end date AND a treatment other than corticosteroid used; - Unresolved with further treatment: any acute rejection with no end date AND a treatment other than corticosteroid used; - Unresolved with no further treatment: any acute rejection with no end date AND ONLY corticosteroid treatment used.
Severity of Biopsy Proven Acute Rejection Episodes | Up to Week 54
  The severity of BPARs is categorized with specific criteria by organ: For kidney transplant participants, according to Banff '97 Diagnostic categories for renal allograft biopsies - Banff '07 update (Acute antibody-mediated rejection I, II, and III, Acute T cell mediated rejection IA, IB, IIA, IIB and III); for liver transplant participants, according to 1997 Banff Schema for grading of Liver Allograft Rejection (mild, moderate, severe or indeterminate/borderline); for heart, according to Standardized Nomenclature of the International Society of Heart and Lung Transplantation (mild, moderate, severe).
Patient survival | Up to Week 54
  Patient survival is defined as the time from first dose of tacrolimus as study drug to the date of death from any cause
Graft survival | Up to Week 54
  Graft survival is defined as the time from the first dose of tacrolimus as study drug to graft loss. Graft loss is defined as retransplantation, nephrectomy (in case of kidney transplantation), death or dialysis (in case of kidney transplantation) ongoing at end of study or at discontinuation, unless superseded by follow-up information.
Efficacy Failure | Up to Week 54
  Efficacy failure is defined as the composite of the following: death, graft loss, BPAR and unknown outcome.
Number of Participants with Adverse Events (Part A) | From first dose of tacrolimus up to 7 days after last dose of tacrolimus prolonged release in Part A (up to 21 days)
  Safety as assessed by adverse events (AEs), which includes abnormalities identified during a medical test (e.g. laboratory tests, vital signs, electrocardiogram, etc.) if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study medication or was clinically significant. A serious AE (SAE) is an event resulting in death, persistent or significant disability/incapacity or congenital anomaly or birth defect, is life-threatening, required or prolonged hospitalization or is considered medically important.
Number of Participants with Adverse Events (Part B) | From first dose of tacrolimus prolonged release in Part A up to 7 days after last dose of tacrolimus prolonged release in Part B (up to 55 weeks)
  Safety as assessed by adverse events (AEs), which includes abnormalities identified during a medical test (e.g. laboratory tests, vital signs, electrocardiogram, etc.) if the abnormality induced clinical signs or symptoms, needed active intervention, interruption or discontinuation of study medication or was clinically significant. A serious AE (SAE) is an event resulting in death, persistent or significant disability/incapacity or congenital anomaly or birth defect, is life-threatening, required or prolonged hospitalization or is considered medically important.

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Europe Ltd.
Locations (16):
- Belgium (2):
  - Site BE21, Brussels
  - Site BE22, Brussels
- Site CZ42, Prague, Czechia
- France (5):
  - Site FR34, Bron
  - Site FR35, Bron
  - Site FR31, Paris
  - Site FR32, Paris
  - Site FR33, Paris
- Site DE41, Heidelberg, Germany
- Italy (2):
  - Site IT74, Bergamo
  - Site IT75, Palermo
- Poland (2):
  - Site PL51, Warsaw
  - Site PL52, Warsaw
- United Kingdom (3):
  - Site GB62, Birmingham
  - Site GB64, London
  - Site GB61, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=216